CLINICAL TRIAL: NCT05482230
Title: Lung Isolation With a Bronchial Blocker Placed in the Lateral Position for Patients Undergoing Thoracic Surgery: a Multicenter, Randomized Clinical Trial
Brief Title: Application of Tracheal Intubation in Lateral Position in Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: xiangming fang (Other)
Collaborators: Red Cross Hospital, Hangzhou, China (Other); The Central Hospital of Lishui City (Other); Affiliated Hospital of Guangdong Medical University (Other); Affiliated Hospital of Jiaxing University (Other); Affiliated Hospital of Shaoxing University (Unknown); Lishui Country People's Hospital (Other)
Responsible Party: Sponsor-Investigator, xiangming fang, Chair Professor, Department of Anesthesiology Vice Dean, School of Medicine and and Pharmaceutical sciences Zhejiang University, First Affiliated Hospital of Zhejiang University
Organization: First Affiliated Hospital of Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2015299
Record Dates: First submitted 2022-07-29; First posted 2022-08-01 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Anesthesia; Tracheal Intubation; Thoracic Surgery
Keywords: Lateral Position; Bronchial occluder
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Intervention Model Description: Intubation and bronchial blocker placement performed in lateral position.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intubation and bronchial blocker placement performed in lateral position (Experimental): In the lateral position group, patients were positioned laterally (as required for surgery) before anesthesia induction. After anesthesia induction, both endotracheal intubation and bronchial blocker placement were performed while the patient remained in the lateral position.
  Interventions: Procedure: Intubation and bronchial blocker placement performed in lateral position
- Intubation and bronchial blocker placement performed in supine position (No Intervention): Intubation and the placement of a bronchial blocker are typically carried out with the patient in the supine position, which is a standard procedure in thoracic surgery.

INTERVENTIONS:
Procedure: Intubation and bronchial blocker placement performed in lateral position — In the lateral position group, patients were positioned laterally (as required for surgery) before anesthesia induction. After anesthesia induction, both endotracheal intubation and bronchial blocker placement were performed while the patient remained in the lateral position.
  Arms: Intubation and bronchial blocker placement performed in lateral position

SUMMARY:
This study investigated the incidence of bronchial blocker malposition in the lateral versus supine position and evaluated the effectiveness of lateral placement.

DETAILED DESCRIPTION:
Routine thoracic surgery anesthesia requires that endotracheal intubation be performed with the patient in the supine position; the patient subsequently needs to be placed in a lateral position through the cooperation of the anesthetist, theatre nurse, and surgeon. Achieving this change in position is time-consuming and likely to result in adverse events, such as loss of the anesthetic airway and arteriovenous catheter, hemodynamic fluctuations, and malposition of the BB which adversely affect anesthesia management and postoperative recovery. For patients with hypertensive heart disease, the risk of cardiovascular and cerebrovascular accidents increases during the perioperative period .

Therefore, we conducted a prospective, randomized, controlled, multi-center study to evaluate the ease, efficacy, and safety of video laryngoscopy-guided intubation and bronchial blocker placement performed in lateral position.

ELIGIBILITY:
The inclusion criteria :

* 80 Years<age ≥18 years;
* American Society of Anesthesiologists (ASA) physical status I-III;
* Undergo thoracic surgery requiring one-lung ventilation.

The exclusion criteria were:

* Risk of difficult intubation based on preoperative assessment (maximum mouth opening <3 cm, body mass index >30 kg/m2, limited neck movement, Mallampati grade IV, or main airway stenosis);
* Right upper bronchus originating at or above the tracheal carina;
* Plan to undergo bronchial sleeve resection, right upper lobectomy, or non-intubated thoracic surgery;
* Evidence or symptoms of acute lung or airway infection;
* History of thoracic surgery;
* Prior thoracic radiotherapy or chemotherapy;
* Preoperative upper extremity pain;
* Severe mental illness or difficulty with communication.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
The incidence of bronchial blocker malposition. | During surgery
  The incidence of bronchial blocker malposition in two groups S and L

SECONDARY OUTCOMES:
The times of bronchial blocker reposition | During surgery
  The times of bronchial blocker reposition in lateral group and supine group
The duration of intubation | During surgery
  The duration of intubation, including the time for single-lumen tube intubation, the time for bronchial blocker placement, and the total intubation time (single-lumen tube intubation plus bronchial blocker placement)
The pressure of ventilation | During surgery
  The pressure of ventilation during mask ventilation, two-lung ventilation (TLV) and one-lung ventilation(OLV)
Intubation-related complications | During surgery, after the patient regained full consciousness and before discharge from the post-anesthesia care unit, on the day after surgery, and 2 weeks postoperatively.
  Intubation-related complications, including airway injury, dental injury, sore throat, and hoarseness
Postural injuries | These complications were assessed at three time points: after the patient regained full consciousness and before discharge from the post-anesthesia care unit, on the day after surgery, and 2 weeks postoperatively.
  Postural injuries were defined as new-onset injuries not present before surgery but occurring within the first 2 weeks postoperatively, including neuropathies, vasculopathies, and musculoskeletal injuries
Lung collapse grade | During surgery
  When the chest wall was opened, the lung collapse was graded as follows: fully collapsed lung, non-collapsed lung with no visible ventilation, or fully ventilated lung
Perioperative vital signs | Immediately after arrival at operating room; Before single lumen tube intubation; After single lumen tube intubation ; One-lung ventilation; Before single lumen tube extubating; 5 minutes after single lumen tube extubating.
  Perioperative vital signs, including mean arterial pressure (MAP), heart rate (HR), and SpO2
Hypoxemia | During surgery
  Hypoxemia was defined as a drop in oxygen saturation (SpO2) below 92%
The satisfaction scores | Perioperative period
  The satisfaction scores of patients, nurses and surgeons. Satisfaction scores were used a 0-10 scale (10 = very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Xiangming Fang, Professor, Principal Investigator — First Affilated Hospital of Zhejiang University
Locations (1):
- Jie Zhao, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
The patient's relevant vital signs and intubation parameters, etc
Supporting Information: Study Protocol

REFERENCES:
- [Background] Almeida C, Freitas MJ, Brandao D, Assuncao JP. [Use of bronchial blocker in emergent thoracotomy in presence of upper airway hemorrhage, and cervical spine fracture: a difficult decision]. Braz J Anesthesiol. 2018 Jul-Aug;68(4):408-411. doi: 10.1016/j.bjan.2017.09.004. Epub 2018 Jan 17. PMID 29342420
- [Background] Lewis JW Jr, Serwin JP, Gabriel FS, Bastanfar M, Jacobsen G. The utility of a double-lumen tube for one-lung ventilation in a variety of noncardiac thoracic surgical procedures. J Cardiothorac Vasc Anesth. 1992 Dec;6(6):705-10. doi: 10.1016/1053-0770(92)90056-d. PMID 1472668
- [Background] Komatsu R, Nagata O, Sessler DI, Ozaki M. The intubating laryngeal mask airway facilitates tracheal intubation in the lateral position. Anesth Analg. 2004 Mar;98(3):858-61, table of contents. doi: 10.1213/01.ane.0000100741.46539.6b. PMID 14980953
- [Background] Goh SY, Thong SY, Chen Y, Kong AS. Efficacy of intubation performed by trainees on patients in the lateral position. Singapore Med J. 2016 Sep;57(9):503-6. doi: 10.11622/smedj.2015165. Epub 2015 Nov 13. PMID 26768062
- [Background] Dimitriou V, Voyagis GS, Iatrou C, Brimacombe J. Flexible lightwand-guided intubation using the intubating laryngeal mask airway in the supine, right, and left lateral positions in healthy patients by experienced users. Anesth Analg. 2003 Mar;96(3):896-898. doi: 10.1213/01.ANE.0000048839.12552.50. PMID 12598281
- [Background] Biswas BK, Agarwal B, Bhattacharyya P, Badhani UK, Bhattarai B. Intubating laryngeal mask for airway management in lateral decubitus state: comparative study of right and left lateral positions. Br J Anaesth. 2005 Nov;95(5):715-8. doi: 10.1093/bja/aei226. Epub 2005 Sep 2. PMID 16143578
- [Background] Takenaka I, Aoyama K, Iwagaki T, Kadoya T. Efficacy of the Airway Scope on tracheal intubation in the lateral position: comparison with the Macintosh laryngoscope. Eur J Anaesthesiol. 2011 Mar;28(3):164-8. doi: 10.1097/EJA.0b013e328340c368. PMID 20962657
- [Background] Jin Y, Ying J, Zhang K, Fang X. Endotracheal intubation under video laryngoscopic guidance during upper gastrointestinal endoscopic surgery in the left lateral position: A randomized controlled trial. Medicine (Baltimore). 2017 Dec;96(52):e9461. doi: 10.1097/MD.0000000000009461. PMID 29384933
- [Background] Li H, Wang W, Lu YP, Wang Y, Chen LH, Lei LP, Fang XM. Evaluation of Endotracheal Intubation with a Flexible Fiberoptic Bronchoscope in Lateral Patient Positioning: A Prospective Randomized Controlled Trial. Chin Med J (Engl). 2016 Sep 5;129(17):2045-9. doi: 10.4103/0366-6999.189069. PMID 27569229
- [Background] Lai HC, Wu ZF. Easier double-lumen tube placement using real-time video laryngoscopy and wireless video fiberoptic bronchoscopy. J Clin Anesth. 2019 Aug;55:132-133. doi: 10.1016/j.jclinane.2018.12.023. Epub 2019 Jan 15. No abstract available. PMID 30658325
- [Background] Birring SS, Brew J, Kilbourn A, Edwards V, Wilson R, Morice AH. Rococo study: a real-world evaluation of an over-the-counter medicine in acute cough (a multicentre, randomised, controlled study). BMJ Open. 2017 Jan 16;7(1):e014112. doi: 10.1136/bmjopen-2016-014112. PMID 28093442
- [Background] Saini S, Bhanot A, Kamal K, Bansal T. An improvised head support to facilitate endotracheal intubation in the lateral position. Acta Anaesthesiol Taiwan. 2015 Sep;53(3):109-11. doi: 10.1016/j.aat.2015.04.001. Epub 2015 Apr 24. No abstract available. PMID 25987271
- [Derived] Li H, Chu L, Ye H, Zhang Y, Li M, Hua Y, Zhang J, Hu H, Wen T, Zhao J, Wan H, Huang L, Lou Y, Tang J, Yan Z, Duan G, Wu J, Wang C, Lu Y, Shen X, Huang C, Song C, Wang Y, Zeng C, Xie G, Fang X. Lung isolation with a bronchial blocker placed in the lateral position for patients undergoing thoracic surgery: A multicenter, randomized clinical trial. J Clin Anesth. 2025 Jun;104:111869. doi: 10.1016/j.jclinane.2025.111869. Epub 2025 May 13. PMID 40367865